CLINICAL TRIAL: NCT04388345
Title: SILENT SINUS SYNDROME (First Case Report, Saudi Arabia With Recommendation)
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Nouf Saloom Alsaloom, Principal Investigator, King Saud University
Other Study IDs: 434200641
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: SILENT SINUS SYNDROME
Keywords: Case report; Silent sinus syndrome; SSS; CT; MRI; Functional endoscopic sinus surgery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Silent sinus syndrome is a rare disorder that presents a diagnostic challenge, most of the patients with this syndrome present with ophthalmological complaints without any nasal sinus symptoms, and it has a painless course and slow development. A case report of a 37-years-old-female who was complaining of severe throbbing pain since 2009, is presented here where the diagnosis of SSS was obtained in 2018, this delay in diagnosing the situation had affected the patient lifestyle tremendously.

DETAILED DESCRIPTION:
Silent sinus syndrome is a rare disorder that presents a diagnostic challenge, most of the patients with this syndrome present with ophthalmological complaints without any nasal sinus symptoms, and it has a painless course and slow development. The syndrome can be diagnosed clinically and confirmed radiologically, and CT imaging is considered the gold standard for its diagnosis. The classical radiographic findings are opacification and collapse of the sinus walls. Functional endoscopic sinus surgery (FESS) is the standard gold treatment of choice to arrest the progression of the disease.

A case report of a 37-years-old-female who was complaining of severe throbbing pain since 2009, is presented here where the diagnosis of SSS was obtained in 2018, this delay in diagnosing the situation had affected the patient lifestyle tremendously.

Accordingly, knowledge of the signs and features of SSS can result in an accurate diagnosis. Suspected cases of silent sinus syndrome require prompt ear, nose, and throat referral for consideration of definitive diagnosis and surgical management. Nasal endoscopy and clinical evaluation are also essential for the diagnosis. Our recommendation is to consider SSS as a differential diagnosis for patients with spontaneous enophthalmos and hypoglobus, even in the absence of maxillary sinus opacification. Moreover, encourage all the specialists in the medical and the dental field to communicate well together in cases like this.

ELIGIBILITY:
Inclusion Criteria:

signs or symptoms in the eyes. signs in the Sinus that seen by X-ray.

Exclusion Criteria:

Children ( <7 years old)

Ages: 37 Years to 37 Years | Sex: Female
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of the signs and features of Silent Sinus Syndeome will result in accurate diagnosis by A computerized tomography (CT) scan. | 10 years
  Suspected cases of silent sinus syndrome require prompt ear, nose and throat referral for consideration of definitive diagnosis and surgical management. Nasal endoscopy and clinical evaluation are essential for the diagnosis, while CT imaging consider the gold standard for its diagnosis. Functional endoscopic sinus surgery is the gold standard treatment to arrest the progression of the disease and the position of the orbital floor can improve following surgical treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cobb AR, Murthy R, Cousin GC, El-Rasheed A, Toma A, Uddin J, Manisali M. Silent sinus syndrome. Br J Oral Maxillofac Surg. 2012 Sep;50(6):e81-5. doi: 10.1016/j.bjoms.2011.10.001. Epub 2011 Nov 1. PMID 22051178
- [Background] Bossolesi P, Autelitano L, Brusati R, Castelnuovo P. The silent sinus syndrome: diagnosis and surgical treatment. Rhinology. 2008 Dec;46(4):308-16. PMID 19146002
- [Background] Guillen DE, Pinargote PM, Guarderas JC. The silent sinus syndrome: protean manifestations of a rare upper respiratory disorder revisited. Clin Mol Allergy. 2013 Dec 9;11(1):5. doi: 10.1186/1476-7961-11-5. PMID 24321328
- [Background] Hourany R, Aygun N, Della Santina CC, Zinreich SJ. Silent sinus syndrome: an acquired condition. AJNR Am J Neuroradiol. 2005 Oct;26(9):2390-2. PMID 16219851
- [Background] Soparkar CN, Patrinely JR, Cuaycong MJ, Dailey RA, Kersten RC, Rubin PA, Linberg JV, Howard GR, Donovan DT, Matoba AY, et al. The silent sinus syndrome. A cause of spontaneous enophthalmos. Ophthalmology. 1994 Apr;101(4):772-8. doi: 10.1016/s0161-6420(94)31267-x. PMID 8152774
- [Background] Vahdani K, Rose GE. Bilateral Silent Sinus (Imploding Antrum) Syndrome. Ophthalmic Plast Reconstr Surg. 2019 May/Jun;35(3):e67-e69. doi: 10.1097/IOP.0000000000001350. PMID 30844910
- [Background] Babar-Craig H, Kayhanian H, De Silva DJ, Rose GE, Lund VJ. Spontaneous silent sinus syndrome (imploding antrum syndrome): case series of 16 patients. Rhinology. 2011 Aug;49(3):315-7. doi: 10.4193/Rhino10.103. PMID 21858262
- [Background] Tribich S, Mahoney CJ, Davies NW. Silent sinus syndrome: an unusual case of facial numbness. Pract Neurol. 2018 Dec;18(6):494-496. doi: 10.1136/practneurol-2017-001807. Epub 2018 Jul 20. PMID 30030411
- [Background] Numa WA, Desai U, Gold DR, Heher KL, Annino DJ. Silent sinus syndrome: a case presentation and comprehensive review of all 84 reported cases. Ann Otol Rhinol Laryngol. 2005 Sep;114(9):688-94. doi: 10.1177/000348940511400906. PMID 16240931
- [Background] Suh JD, Ramakrishnan V, Lee JY, Chiu AG. Bilateral silent sinus syndrome. Ear Nose Throat J. 2012 Dec;91(12):E19-21. doi: 10.1177/014556131209101217. PMID 23288826